CLINICAL TRIAL: NCT03802227
Title: A Phase 1 Double-Blind, Double-Dummy, Parallel-Group, Randomized, Positive Control Study Using fMRI to Evaluate the Effect of NKTR-181 on Brain Activity in Healthy, Non-physically Dependent Recreational Opioid Users
Brief Title: A Study Using fMRI Imaging to Evaluate the Effect of NKTR-181 on Brain Activity in Healthy, Non-physically Dependent Recreational Opioid Users.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 18-181-26
Record Dates: First submitted 2018-11-15; First posted 2019-01-14 (Actual); Results first posted 2021-05-27 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Moderate to Severe Chronic Pain
MeSH Terms: interventions — NKTR-181

STUDY DESIGN:
Intervention Model Description: A double-blind, double-dummy, parallel-group, randomized, positive control study.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): NKTR-181 400 mg and oxycodone IR placebo
  Interventions: Drug: NKTR-181
- Group 2 (Experimental): Oxycodone IR 40 mg and NKTR-181 placebo
  Interventions: Drug: Oxycodone IR

INTERVENTIONS:
Drug: NKTR-181 — A combination of NKTR-181 and oxycodone IR placebo
  Arms: Group 1
Drug: Oxycodone IR — A combination of oxycodone IR and NKTR-181 placebo
  Arms: Group 2

SUMMARY:
The main purpose of this study is to evaluate the effect of NKTR-181 on brain activity in healthy, non-physically dependent recreational opioid users. This study will last about 88 days for each participant.

DETAILED DESCRIPTION:
This study is a single-center study in which approximately 24 subjects will be randomized to one of two treatment groups. Subjects will enter a screening period between Day -28 and Day -2. Upon meeting all criteria for enrollment, on Day -1 subjects will enter the clinical research study unit (CRSU) for an overnight confinement. On Day 1, subjects will undergo a baseline MRI and will then be randomized to NKTR-181 or oxycodone immediate release (IR). Once randomized, subjects will receive a single dose of study drug (NKTR-181 or oxycodone IR) and matched alternate-treatment placebo. Subjects will undergo a series of three fMRIs (functional magnetic resonance imaging) post dose (at hours 1, 2, and 4). At post-dose hours 0.5, 1, 2, 3, 4, 5, 6, and 8, pupillometry will be performed and PK blood samples will be drawn. Following a 14- to 17-day safety follow-up period, subjects will return to the research facility clinic for the End of Study (EOS) visit (Day 16-19).

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy male and female recreational opioid users, 18-65 years of age inclusive.
* Body Mass Index (BMI) between 19.0 to 45.0kg/m2
* Have at least one urine drug screen positive for opioids during Screening to confirm recreational opioid use. Subjects testing positive for methadone or buprenorphine prescribed for treatment will be excluded.
* Subjects must agree to practice adequate contraception as outlined in the protocol.

Key Exclusion Criteria:

* Any metal fragments or other bodily metal that would pose a risk to subjects during MRI scanning as determined by the MRI technologist and/or MRI physicist
* Any clinically significant disease or condition that might compromise the cardiovascular, hematological, renal, hepatic, pulmonary, endocrine, central nervous, or gastrointestinal systems or other conditions that may interfere with the absorption, distribution, metabolism, or excretion of the study drug or would place the subject at increased risk
* History of clinically significant acute asthma or other obstructive airway disease requiring daily controller medication or any condition that may increase the risk for respiratory depression
* Current neurologic conditions such as convulsive disorders, or history of severe head injury.
* Any current DSM-5 axis I psychiatric disorder or neurological disorder requiring ongoing treatment
* Current substance use disorder (moderate to severe), other than Opioid, Nicotine, THC (tetrahydrocannabinol), cocaine, or caffeine as defined by DSM-5
* Physical dependence of opioids
* History of claustrophobia or any other psychiatric disorder that would preclude subject tolerance of MRI procedures.
* Current use of any medication that could affect central nervous system blood flow (e.g. certain cardiovascular medications, triptan migraine medications)
* Clinical Opiate Withdrawal Scale (COWS) score of greater than 5 during screening or prior to first scan.
* Positive urine drug screen for buprenorphine or methadone immediately prior to the first scan.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2020-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (1):
- Investigator Site - Richmond, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Treatment assignments were based on a computer-generated randomization scheduled prepared by SynteractHCR Inc. prior to study start
Groups:
- NKTR-181: Two 200 mg NKTR-181 tablets and 1 placebo capsule for oxycodone IR
- Oxycodone IR 40 mg: Once capsule of Oxycodone IR 40 mg and 2 placebo tablets for NKTR-181
Period: Overall Study
Arm/Group | NKTR-181 | Oxycodone IR 40 mg
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- NKTR-181: Two 200 mg NKTR-181 tablets and 1 placebo capsule for oxycodone IR oxycodone IR
- Oxycodone IR 40 mg: One capsule of Oxycodone IR 40 mg and 2 placebo tablets for NKTR-181
- Total: Total of all reporting groups
Arm/Group | NKTR-181 | Oxycodone IR 40 mg | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (7.42) | 43.5 (3.42) | 41.0 (5.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height (cm) [Mean (Standard Deviation); unit: centimeters] | 166.3 (5.94) | 182.0 (2.44) | 174.1 (9.39)
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 81.5 (21.30) | 83.8 (5.93) | 82.7 (14.52)
BMI (kg/m2) [Mean (Standard Deviation); unit: kilograms per meter squared] | 29.7 (8.83) | 25.3 (2.12) | 27.5 (6.39)
Systolic Blood Pressure (mm Hg) [Mean (Standard Deviation); unit: millimeters of Hg] | 143.5 (11.47) | 127.3 (12.74) | 135.4 (14.19)
Diastolic Blood Pressure (mm Hg) [Mean (Standard Deviation); unit: millimeters of Hg] | 91.3 (18.63) | 74.5 (12.66) | 82.9 (17.25)
Pulse Rate (bpm) [Mean (Standard Deviation); unit: beats per minute] | 74.5 (6.40) | 74.3 (4.35) | 74.4 (5.07)
Respiratory Rate (breaths per minute) [Mean (Standard Deviation); unit: breaths per minute] | 14.0 (2.31) | 17.5 (1.00) | 15.8 (2.49)
SpO2 (%) [Mean (Standard Deviation); unit: %] | 97.3 (0.96) | 97.5 (1.91) | 97.4 (1.41)
Temperature (degrees Celsius) [Mean (Standard Deviation); unit: degrees Celsius] | 36.7 (0.37) | 36.8 (0.27) | 36.7 (0.30)

OUTCOME MEASURES:

1. Primary Outcome: Brain Activity Measured Via fMRI
Description: The primary objective of the study was to evaluate the effects of NKTR-181 on brain activity. Functional MRI assessments in subjects administered opioids such as morphine, buprenorphine, and nalbuphine have shown drug-induced signaling changes in reward structures such as the nucleus accumbens, orbitofrontal cortex, and hippocampus, as well as changes in the functional connectivity of reward circuitry (Becerra, 2006; Gear, 2013; Upadhyay, 2012).
Time Frame: 8 hour period following dose of NKTR-181
Population: Subjects who had sufficient MRI data for NKTR-181 or oxycodone IR treatment to allow for analysis of modulation of brain circuitry.
Measure: Mean (Standard Deviation); unit: Correlation Coefficient
Arm/Group | NKTR-181 | Oxycodone IR 40 mg
Number analyzed (Participants) | 4 | 4
Correlation Coefficient
  Effective Connectivity between ACC and R Hippocampus at Baseline | 0.0 (0.12) | 0.2 (0.34)
  Effective Connectivity between ACC and R Hippocampus after 1 hour | 0.0 (0.28) | 0.0 (0.21)
  Effective Connectivity between ACC and R Hippocampus after 2 hours | 0.1 (0.20) | -0.1 (0.10)
  Effective Connectivity between ACC and R Hippocampus after 4 hours | 0.0 (0.20) | 0.0 (0.48)
  Effective Connectivity between ACC and R Hippocampus after 8 hours: number analyzed (Participants) | 2 | 3
  Effective Connectivity between ACC and R Hippocampus after 8 hours | -0.1 (0.02) | 0.2 (0.07)
  Effective Connectivity between R Amygdala and mPFC at Baseline | 0.1 (0.38) | 0.0 (0.14)
  Effective Connectivity between R Amygdala and mPFC after 1 hour | -0.2 (0.41) | 0.1 (0.34)
  Effective Connectivity between R Amygdala and mPFC after 2 hours | 0.2 (0.21) | 0.4 (0.51)
  Effective Connectivity between R Amygdala and mPFC after 4 hours | 0.2 (0.26) | 0.1 (0.21)
  Effective Connectivity between R Amygdala and mPFC after 8 hours: number analyzed (Participants) | 2 | 3
  Effective Connectivity between R Amygdala and mPFC after 8 hours | 0.1 (0.54) | 0.1 (0.18)

2. Secondary Outcome: Change in Pupil Diameter Via Pupillometry
Description: Analysis of change in pupil diameter after administration of NKTR-181 or Oxycodone IR.
Time Frame: 24 hour period following dose administration Day 1 to 2
Population: Subjects who received at least one dose of NKTR-181 or oxycodone IR and did not have unexpected pupillary dilation as a result of technical issues during the procedure.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | NKTR-181 | Oxycodone IR 40 mg
Number analyzed (Participants) | 4 | 4
millimeters
  Baseline Pupil Diameter | 4.45 (1.198) | 4.81 (1.717)
  Pupil Diameter After 1 Hour: number analyzed (Participants) | 3 | 3
  Pupil Diameter After 1 Hour | 5.03 (0.443) | 4.87 (1.624)
  Pupil Diameter After 2 Hours | 4.82 (1.550) | 4.97 (1.747)
  Pupil Diameter After 4 Hours | 4.34 (0.985) | 5.32 (1.723)
  Pupil Diameter After 6 Hours: number analyzed (Participants) | 2 | 4
  Pupil Diameter After 6 Hours | 3.99 (2.213) | 5.01 (1.086)
  Pupil Diameter After 8 Hours: number analyzed (Participants) | 3 | 2
  Pupil Diameter After 8 Hours | 4.28 (1.161) | 5.07 (1.115)
  Pupil Diameter After 12 Hours: number analyzed (Participants) | 1 | 1
  Pupil Diameter After 12 Hours | 4.91 (NA) — There is only one participant | 3.87 (NA) — There is only one participant
  Pupil Diameter After 24 Hours: number analyzed (Participants) | 2 | 2
  Pupil Diameter After 24 Hours | 4.61 (0.403) | 4.20 (0.191)

3. Secondary Outcome: Plasma Drug Concentration
Description: Plasma drug concentration for NKTR-181 and Oxycodone IR over 24 hours.
Time Frame: 24 hour period following dose administration Day 1 to 2
Population: Consisted of all subjects who had sufficient plasma concentration data to facilitate the calculation of maximum plasma drug concentration as determined by the pharmacokineticist.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | NKTR-181 | Oxycodone IR 40 mg
Number analyzed (Participants) | 4 | 4
ng/mL
  Plasma Drug Concentration at Hour 1 | 1970 (477) | 35.7 (33.9)
  Plasma Drug Concentration at Hour 2 | 2360 (1230) | 54.1 (13.1)
  Plasma Drug Concentration at Hour 4: number analyzed (Participants) | 4 | 3
  Plasma Drug Concentration at Hour 4 | 1350 (656) | 46.7 (15.3)
  Plasma Drug Concentration at Hour 8: number analyzed (Participants) | 2 | 2
  Plasma Drug Concentration at Hour 8 | 388 (230) | 27.1 (7.47)
  Plasma Drug Concentration at Hour 12: number analyzed (Participants) | 2 | 1
  Plasma Drug Concentration at Hour 12 | 185 (30.4) | 14.8 (NA) — Only one sample was collected for this measurement
  Plasma Drug Concentration at Hour 24: number analyzed (Participants) | 2 | 1
  Plasma Drug Concentration at Hour 24 | 63.5 (13.7) | 3.9 (NA) — Only one sample was collected for this measurement

4. Secondary Outcome: Time to Maximum Concentration (Tmax)
Description: The amount of time needed for maximum drug concentration to be reached.
Time Frame: 24 hour period following dose administration Day 1 to 2
Population: Consisted of all subjects who had sufficient plasma concentration data to facilitate the calculation of the time to maximum plasma drug concentration as determined by the pharmacokineticist.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | NKTR-181 | Oxycodone IR 40 mg
Number analyzed (Participants) | 4 | 4
ng/mL
  Plasma Drug Concentration at Hour 1 | 1970 (477) | 35.7 (33.9)
  Plasma Drug Concentration at Hour 2 | 2360 (1230) | 54.1 (13.1)
  Plasma Drug Concentration at Hour 4: number analyzed (Participants) | 4 | 3
  Plasma Drug Concentration at Hour 4 | 1350 (656) | 46.7 (15.3)
  Plasma Drug Concentration at Hour 8: number analyzed (Participants) | 2 | 2
  Plasma Drug Concentration at Hour 8 | 388 (230) | 27.1 (7.47)
  Plasma Drug Concentration at Hour 12: number analyzed (Participants) | 2 | 1
  Plasma Drug Concentration at Hour 12 | 185 (30.4) | 14.8 (NA) — There is only one participant
  Plasma Drug Concentration at Hour 24: number analyzed (Participants) | 4 | 1
  Plasma Drug Concentration at Hour 24 | 63.5 (13.7) | 3.9 (NA) — There is only one participant
  Time to Maximum Concentration (Tmax) measured in hours | 1.54 (0.676) | 2.21 (1.02)

5. Secondary Outcome: Treatment-Emergent Adverse Events (TEAEs)
Description: Number of patients who experienced any type of adverse event as a result of one of the treatments.
Time Frame: 19 days
Population: Consisted of all subjects who received at least 1 dose of NKTR-181 or Oxycodone IR.
Measure: Count of Participants; unit: Participants
Groups:
- NKTR-181: NKTR-181 400 mg and placebo for oxycodone IR one tablet of each once
- Oxycodone IR 40 mg: Oxycodone IR 40 mg and placebo for NKTR-181 one tablet of each once
Arm/Group | NKTR-181 | Oxycodone IR 40 mg
Number analyzed (Participants) | 4 | 4
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 19 days post-dose of NKTR-181 or Oxycodone IR 40 mg
Description: All adverse events and their duration were listed. Adverse events that occurred on or after study dose administration were summarized. Verbatim terms were mapped to PTs and system organ classes (SOC) using the Medical Dictionary for Regulatory Activities (MedDRA).
Arm/Group | NKTR-181 | Oxycodone IR 40 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/4 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NKTR-181 (N=4) | Oxycodone IR 40 mg (N=4)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — One subject experienced back pain that was treated with paracetamol and resolved within 1-2 days. The back pain was deemed not related to the study drug (NKTR-181).
Insomnia (General disorders) | 1 (1) | 0 (0) — One subject experienced insomnia that was treated with trazodone and resolved within 1-2 days. The insomnia was deemed not related to the study drug (NKTR-181)

LIMITATIONS AND CAVEATS:
The study was originally planned for 24 patients. However enrollment was stopped due to the CDP being stopped at 8 and therefore limits the generalizability of this data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are restrictions to the PI's rights to discuss or publish trial results.

DOCUMENTS (2):
  • Study Protocol (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/27/NCT03802227/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT03802227/SAP_001.pdf